CLINICAL TRIAL: NCT04913181
Title: Application of Artificial Intelligence Sepsis Prediction Model to Assist ICU Clinical Decision
Brief Title: Artificial Intelligence for Sepsis Prediction in ICU
Acronym: AICUSepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: SHZJU-ICU2020-202
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Artificial Intelligence; Septic Shock; Intensive Care Unit Psychosis
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis prediction model: This group of people was used for the clinician's decision, and the sepsis prediction model was used simultaneously for the prediction, but the model was not involved in the decision, and was only used for verification
  Interventions: Diagnostic Test: Artificial intelligence sepsis prediction model
- Daily clinical judgment of doctors: This group of people was used for the clinician's decision without sepsis prediction model.
  Interventions: Diagnostic Test: Artificial intelligence sepsis prediction model

INTERVENTIONS:
Diagnostic Test: Artificial intelligence sepsis prediction model — The main purpose of this paper is to evaluate the accuracy of the sepsis prediction model established in the early stage. The occurrence of sepsis is determined by the daily clinical judgment of doctors, and the results of sepsis prediction model are matched and corrected.

SUMMARY:
The development of sepsis prediction model in line with Chinese population, and extended to clinical, assist clinicians for early identification, early intervention, has a good application prospect. This study is a prospective observational study, mainly to evaluate the accuracy of the previously established sepsis prediction model. The occurrence of sepsis was determined by doctors' daily clinical judgment, and the results of the sepsis prediction model were matched and corrected to improve the clinical accuracy and applicability of the sepsis prediction model.

DETAILED DESCRIPTION:
The sepsis prediction model adopted in this study has been completed in the preliminary preparation, which was constructed on 7,000 patients since the establishment of comprehensive ICU, and the sepsis 3.0 diagnostic standard was adopted.The sepsis prediction model was built using Python platform and XGBoost algorithm, which was used to predict the incidence of sepsis in ICU patients within 24 hours. The overall accuracy was 82%, and the area under the Auroc curve was 0.854.

Patients who met the inclusion and exclusion criteria were given a daily prediction of sepsis model, and a quantitative checklist was formed based on the test results.There are two kinds of forecast outcomes: low risk and high risk.Quantitative checklists are available to attending physicians to improve diagnostic efficiency.The results were kept confidential to the clinician.

All patients were diagnosed with sepsis by two senior attending physicians at a fixed time. The diagnosis consisted of two types: yes and no.If two attending physicians have different opinions, the third attending physician will be included for correction diagnosis, and the presence of sepsis will be determined in a 2:1 manner.The attending physicians are independent of each other.

When the diagnosis results of the attending physician are input into the system, the prediction results of yesterday's sepsis prediction model are compared and calculated to determine the accuracy of the prediction model

ELIGIBILITY:
Inclusion Criteria:

All patients with acute critical illness who are eligible for admission to ICU during the study period

Exclusion Criteria:

1. Patients under the age of 16;
2. Pregnant and parturient women;
3. Patients who planned to be admitted to the department for surgery and transferred the next day after evaluation;
4. Patients admitted to the department and diagnosed with sepsis;
5. Patients with ICU stay less than 24 hours;

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who met the inclusion and exclusion criteria were predicted daily by sepsis model, and a quantitative list was formed according to the test results. There are two kinds of prediction results: low risk and high risk. The quantitative list is open to attending physicians to improve the efficiency of diagnosis. The predicted results are kept secret from clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of model diagnosis | 2 years
  Evaluation of the accuracy of prediction model in clinical application

IPD SHARING:
Plan to Share IPD: No